CLINICAL TRIAL: NCT03606941
Title: Effect of Electroacupuncture on the Incidence of Postoperative Delirium in Elderly Patients Undergoing the Major Surgery：a Prospective, Multicenter, Double-blind, Randomized Controlled Trial
Brief Title: Effect of Electroacupuncture on the Incidence of Postoperative Delirium in Elderly Patients Undergoing the Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Department of Anesthesiology, Director, Chief physician, Professor, Doctoral tutor, Tianjin Nankai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NKYY_YX_IRB_2017_036_02
Record Dates: First submitted 2018-07-02; First posted 2018-07-31 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Delirium
Keywords: electroacupuncture; delirium; the elderly; surgery, major
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture treatment (Experimental): Participants in the treatment group received acupuncture (0.30mm×70mm) at bilaterally Shenmen (HT7) acupoints (0.3-0.5 inch), Neiguan (PC6) acupoints (0.5-1 inch), Baihui (DU20) acupoint (0.5-0.8 inch) and Yintang (EX-HN3) acupoint (0.3-0.5 inch) 30 minutes before anesthesia induction. After "Deqi", electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China) is connected and maintained the end of operation.
  Interventions: Device: electroacupuncture treatment
- sham electroacupuncture treatment (Sham Comparator): Participants in the control group received shallow needling (0.30mm×25mm) at bilateral sham HT7, PC6, DU20 and EX-HN3 (nonacupoints located 1 inch beside acupoints, about 20mm). Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output.
  Interventions: Device: sham electroacupuncture treatment

INTERVENTIONS:
Device: electroacupuncture treatment — Participants in the electroacupuncture group received acupuncture (0.30mm×70mm) at bilaterally Shenmen (HT7) acupoints (0.3-0.5 inch), Neiguan (PC6) acupoints (0.5-1 inch), Baihui (DU20) acupoint (0.5-0.8 inch) and Yintang (EX-HN3) acupoint (0.3-0.5 inch) 30 minutes before anesthesia induction. After "Deqi", electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China) is connected with the density wave (2/100 Hz), width 0.25 ms, intensity of 1 ~ 30 mA (gradually increase to the patient's maximum tolerance) and maintained the end of operation.
  Arms: electroacupuncture treatment
Device: sham electroacupuncture treatment — Participants in the sham electroacupuncture group received shallow needling (0.30mm×25mm) at bilateral sham HT7, PC6, DU20 and EX-HN3 (nonacupoints located 1 inch beside acupoints, about 20mm). Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output, and retained the needle until the end of surgery.
  Arms: sham electroacupuncture treatment

SUMMARY:
1. Title: Effect of electroacupuncture on the incidence of postoperative delirium in elderly patients undergoing the major surgery.
2. Research center: Multicenter
3. The Design of the study: Randomized, double-blind, controlled study
4. The population of the study: Elderly patients（65≤age<90 years），it is planned to select a period/time limit for gastrointestinal tumor surgery, bile duct surgery, thoracic surgery or orthopedic surgery and so on under general anesthesia, and the estimated operation time≥ 2 hours.
5. Sample size: Enroll 1100 patients (550 patients in each group)
6. Interventions: Participants in the treatment group received acupuncture (0.30mm×70mm) at bilaterally Shenmen (HT7) acupoints (0.3-0.5 inch), Neiguan (PC6) acupoints (0.5-1 inch), Baihui (DU20) acupoint (0.5-0.8 inch) and Yintang (EX-HN3) acupoint (0.3-0.5 inch) 30 minutes before anesthesia induction. After "Deqi", electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China) is connected and maintained the end of operation. Participants in the control group received shallow needling (0.30mm×25mm) at bilateral sham HT7, PC6, DU20 and EX-HN3 (nonacupoints located 1 inch beside acupoints, about 20mm). Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output.
7. The aim of the research: To investigate the effect of electroacupuncture on the incidence of postoperative delirium within 5 days in elderly patients undergoing the major surgery.
8. Outcome： 1) Primary outcome：The incidence of delirium within 5 days after surgery；The effects on postoperative NRS pain and sleep quality scores； 2)Secondary outcome：Duration of mechanical ventilation in patients with endotracheal intubation on ICU admission; Length of stay in ICU and Length of stay in hospital after surgery; Incidence of postoperative complications (including re-hospitalization); 30-day life quality and cognitive function after surgery; All-cause 30-day mortality after surgery.
9. The estimated duration of the study：3-4 years.

DETAILED DESCRIPTION:
This study is a large sample, randomized, double-blinded, placebo-controlled and long-term follow-up design. In this study, bilateral Shenmen, Neiguan, Baihui and Yintang acupoints were selected for perioperative electroacupuncture treatment, accompanied with evaluating the incidence of delirium within 5 days after surgery,the effects on postoperative NRS pain and sleep quality scores as well as the detection of blood biochemical indexes such as serum S100β, brain derived neurotrophic factor (BDNF), interleukin-6 and interleukin-8. To clarify the effect of electroacupuncture on the incidence of postoperative delirium in elderly patients undergoing the major surgery is of great significance to the clinical applications and popularization of traditional acupuncture treatment perioperatively across the world.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥65 and <90 years old；
2. Planning to undergo select timed/limited surgery such as gastrointestinal tumor surgery, bile duct surgery and thoracic surgery etc under general anesthesia, and the estimated operation time is more than 2 hours;；
3. Treatment without radiotherapy or chemotherapy prior to surgery；
4. Agree to participate in this study and sign informed consent；

Exclusion Criteria:

1. Refuse to participate in this study；
2. Preoperative history of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis；
3. Inability to communicate in the preoperative period to complete preoperative evaluation because of severe dementia, coma, language barrier；
4. Brain injury or neurosurgery；
5. Critical condition (if the ASA grade is greater than or equal to grade IV before surgery); Severe renal impairment (dialysis treatment before surgery); Severe liver function impairment (Child-Pugh level C); Preoperative combined with severe heart disease, LVEF < 30%;
6. Previous experience of acupoint stimulation therapy or non-insensitive to acupoint stimulation；
7. The attending physician or researcher considers that there are other circumstances (reasons to be noted) that are not suitable for participation in this study.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The incidence of delirium within 5 days after surgery | an average of one year
  Using confusion assessment method (CAM) or CAM-ICU methods to assess delirium

SECONDARY OUTCOMES:
Duration of mechanical ventilation in patients with endotracheal intubation on ICU | an average of 1 year
  Duration of mechanical ventilation and endotracheal intubation in ICU
Length of stay in hospital after surgery | 12 months
  postoperative ICU stay time and hospitalization time
Incidence of non-delirium complications during the first 30 days after surgery (including re-hospitalization) | up to 1 year
  cardiac events, cerebrovascular events, renal injury, infections, etc
All-cause 30-day mortality after surgery | 1 year
  All reasons (such as infection, hemorrhage) caused the mortality during the first 30 days after surgery
The effects on postoperative pain scores | up to 12 months
  NRS method is used to evaluate the pain scores of patients (0 points to complete Painless, 10 points to the maximum pain that can be tolerated)
The effects on postoperative sleep quality scores | up to one year
  Using the NRS method (0 for the best quality of sleep and 10 for the worst quality of sleep)

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, MD,PhD, Study Chair — Tianjin Nankai Hospital
Locations (1):
- Electroacupuncture Apparatus, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oh ES, Fong TG, Hshieh TT, Inouye SK. Delirium in Older Persons: Advances in Diagnosis and Treatment. JAMA. 2017 Sep 26;318(12):1161-1174. doi: 10.1001/jama.2017.12067. PMID 28973626
- [Result] Robinson TN, Raeburn CD, Tran ZV, Angles EM, Brenner LA, Moss M. Postoperative delirium in the elderly: risk factors and outcomes. Ann Surg. 2009 Jan;249(1):173-8. doi: 10.1097/SLA.0b013e31818e4776. PMID 19106695
- [Result] Naeije G, Pepersack T. Delirium in elderly people. Lancet. 2014 Jun 14;383(9934):2044-2045. doi: 10.1016/S0140-6736(14)60993-4. No abstract available. PMID 24931688
- [Result] Morandi A, Jackson JC. Delirium in the intensive care unit: a review. Neurol Clin. 2011 Nov;29(4):749-63. doi: 10.1016/j.ncl.2011.08.004. PMID 22032658
- [Result] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Result] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Result] Inouye SK, Schlesinger MJ, Lydon TJ. Delirium: a symptom of how hospital care is failing older persons and a window to improve quality of hospital care. Am J Med. 1999 May;106(5):565-73. doi: 10.1016/s0002-9343(99)00070-4. PMID 10335730
- [Result] Franco K, Litaker D, Locala J, Bronson D. The cost of delirium in the surgical patient. Psychosomatics. 2001 Jan-Feb;42(1):68-73. doi: 10.1176/appi.psy.42.1.68. PMID 11161124
- [Result] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Result] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Result] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Result] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Result] Avidan MS, Maybrier HR, Abdallah AB, Jacobsohn E, Vlisides PE, Pryor KO, Veselis RA, Grocott HP, Emmert DA, Rogers EM, Downey RJ, Yulico H, Noh GJ, Lee YH, Waszynski CM, Arya VK, Pagel PS, Hudetz JA, Muench MR, Fritz BA, Waberski W, Inouye SK, Mashour GA; PODCAST Research Group. Intraoperative ketamine for prevention of postoperative delirium or pain after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Lancet. 2017 Jul 15;390(10091):267-275. doi: 10.1016/S0140-6736(17)31467-8. Epub 2017 May 30. PMID 28576285
- [Result] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Result] Sieber FE. Postoperative delirium in the elderly surgical patient. Anesthesiol Clin. 2009 Sep;27(3):451-64, table of contents. doi: 10.1016/j.anclin.2009.07.009. PMID 19825486
- [Result] Avramescu S, Wang DS, Choi S, Orser BA. Preventing delirium: beyond dexmedetomidine. Lancet. 2017 Mar 11;389(10073):1009. doi: 10.1016/S0140-6736(17)30661-X. No abstract available. PMID 28290991
- [Result] Lin JG, Chen YH. The mechanistic studies of acupuncture and moxibustion in Taiwan. Chin J Integr Med. 2011 Mar;17(3):177-86. doi: 10.1007/s11655-011-0664-8. PMID 21359918
- [Result] Chernyak GV, Sessler DI. Perioperative acupuncture and related techniques. Anesthesiology. 2005 May;102(5):1031-49; quiz 1077-8. doi: 10.1097/00000542-200505000-00024. PMID 15851892
- [Result] Liu Z, Liu Y, Xu H, He L, Chen Y, Fu L, Li N, Lu Y, Su T, Sun J, Wang J, Yue Z, Zhang W, Zhao J, Zhou Z, Wu J, Zhou K, Ai Y, Zhou J, Pang R, Wang Y, Qin Z, Yan S, Li H, Luo L, Liu B. Effect of Electroacupuncture on Urinary Leakage Among Women With Stress Urinary Incontinence: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2493-2501. doi: 10.1001/jama.2017.7220. PMID 28655016
- [Result] Vickers AJ, Linde K. Acupuncture for chronic pain. JAMA. 2014 Mar 5;311(9):955-6. doi: 10.1001/jama.2013.285478. PMID 24595780
- [Result] Liu Z, Yan S, Wu J, He L, Li N, Dong G, Fang J, Fu W, Fu L, Sun J, Wang L, Wang S, Yang J, Zhang H, Zhang J, Zhao J, Zhou W, Zhou Z, Ai Y, Zhou K, Liu J, Xu H, Cai Y, Liu B. Acupuncture for Chronic Severe Functional Constipation: A Randomized Trial. Ann Intern Med. 2016 Dec 6;165(11):761-769. doi: 10.7326/M15-3118. Epub 2016 Sep 13. PMID 27618593
- [Result] Lin R, Li X, Liu W, Chen W, Yu K, Zhao C, Huang J, Yang S, Peng H, Tao J, Chen L. Electro-acupuncture ameliorates cognitive impairment via improvement of brain-derived neurotropic factor-mediated hippocampal synaptic plasticity in cerebral ischemia-reperfusion injured rats. Exp Ther Med. 2017 Sep;14(3):2373-2379. doi: 10.3892/etm.2017.4750. Epub 2017 Jul 10. PMID 28962170
- [Result] Zhang Q, Li YN, Guo YY, Yin CP, Gao F, Xin X, Huo SP, Wang XL, Wang QJ. Effects of preconditioning of electro-acupuncture on postoperative cognitive dysfunction in elderly: A prospective, randomized, controlled trial. Medicine (Baltimore). 2017 Jun;96(26):e7375. doi: 10.1097/MD.0000000000007375. PMID 28658163
- [Result] Matsumoto-Miyazaki J, Ushikoshi H, Miyata S, Miyazaki N, Nawa T, Okada H, Ojio S, Ogura S, Minatoguchi S. Acupuncture and Traditional Herbal Medicine Therapy Prevent Deliriumin Patients with Cardiovascular Disease in Intensive Care Units. Am J Chin Med. 2017;45(2):255-268. doi: 10.1142/S0192415X17500161. Epub 2017 Feb 23. PMID 28231740